CLINICAL TRIAL: NCT02197845
Title: Enhancing Use of Hydroxyurea In Sickle Cell Disease Using Patient Navigators
Acronym: SHiP HU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eastern Virginia Medical School (Other); Children's Hospital of The King's Daughters (Other); Virginia Department of Health (Other Government); James Madison University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HM14641; 1R18HL112737-01 (NIH)
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; hydroxyurea; patient navigator; community health worker; public health worker; fetal hemoglobin; health services research
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia | interventions — Patient Navigation; Community Health Workers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Phase I: Recruitment into Specialty Care (Experimental): Participants in the Phase I Experimental Arm are enrolled into SCD specialty care. PN's will contact patient up to 3 times to assure patients have had an initial visit by 3 months time.
  Interventions: Behavioral: Recruitment into Specialty Care
- Phase II: Patient Navigator Arm (Experimental): Participants in the Phase II Experimental Arm follow routine clinical care and are assigned a Patient Navigator. A specially trained (SCD specefic)PN will work with participants for one year. Participants will be contacted by their Navigator weekly for the first 6 months, then biweekly for the second 6 months.
  Interventions: Behavioral: Patient Navigator
- Phase II: Passenger Arm (No Intervention): No Intervention. Participants in the Phase II Passenger Arm follow routine clinical care.

INTERVENTIONS:
Behavioral: Patient Navigator — A specially trained (SCD knowledgable) Patient Navigator will act as a liaison who assists participants in increasing adherence to HU through disease education, addressing barriers to care and improving adherence to HU. PN utilize various techniques geared toward the individual patients needs. Interventions utilized by a PN include improving disease management skills, educational materials about disease, HU adherence, motivational interviewing, care coordination and social support.
  Other Names: Public Health Worker; Community Health Worker
  Arms: Phase II: Patient Navigator Arm
Behavioral: Recruitment into Specialty Care — A specially trained (SCD knowledgeable) Patient Navigator will act as a liaison to participants in increasing adherence to Hydroxyurea. Interventions utilized by a PN include teaching disease management skills, addressing barriers to care, disease education, HU management, motivational interviewing, care coordination and social support.
  Other Names: Sickle Cell Disease Specialty Care
  Arms: Phase I: Recruitment into Specialty Care

SUMMARY:
Multi-phase, patient navigator-based program in the Richmond and Tidewater regions of Virginia to demonstrate:

1. the feasibility of using patient navigators to improve the percentage of children and adult (age 15 and older) patients with sickle cell disease (SCD) in SCD specialty care
2. the efficacy of using patient navigators to improve hydroxyurea (HU) (re-)initiation and adherence among adult patients with SCD eligible for HU

(Patient navigators may also be known as public health workers.)

DETAILED DESCRIPTION:
The state of Virginia, including the Virginia Department of Health and three academic medical centers and one federally qualified health center, plans a two-phase demonstration, first of improvement in the percentage of adults with SCD who are in SCD specialty care (Phase I), then of improvement in adherence to HU of eligible SCD adults (Phase II). Both phases will use existing academic SCD providers, and an innovative, multimodal strategy, featuring specially trained SCD patient navigators (PNs), that addresses barriers to care and to HU use. In Phase I we will demonstrate the feasibility of utilizing PNs to overcome patient access barriers to SCD care. In Phase II we will test the efficacy of PNs for overcoming barriers to acceptance of and adherence with HU therapy. Patients will be randomized to a PN arm or to a usual care arm. Providers will implement NIH guidelines for HU eligibility and prescribing in both arms. All HU eligible patients will be offered HU at each clinical visit. Among patients prescribed HU, if a maximum tolerated dose (MTD, defined in end points) has not been reached, providers will dose escalate every 8-12 weeks to MTD, rather than to clinical effect, before declaring treatment success or failure.

This project will be critically important and impactful by demonstrating the feasibility of a statewide community-based strategy to assist vulnerable SCD adults in obtaining SCD specialty care and likely prolonging life, a model that other states could adopt.

ELIGIBILITY:
PHASE I:

Inclusion Criteria:

* Patient Self Report of Sickle Cell Disease (Genotypes: Hb SS, SC, SBoThal, SB+Thal)
* 15 years or older
* Virginia resident

Exclusion Criteria:

-Visited one of a pre-selected list of sickle cell specialists in Virginia within the last 6 months

PHASE II:

Inclusion Criteria:

* Sickle Cell Disease (SCD) patient (Genotypes: SS or SBoThal)
* Eligible for Hydroxyurea (according to NIH guidelines)
* 15 years or older
* Virginia resident

Exclusion Criteria:

* Pregnancy
* Enrollment in scheduled chronic transfusion program
* SCD Genotype: Hb SC and SB+Thal)

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Phase I: Percent of enrolled Phase I subjects who complete a provider visit by 3 months post enrollment | 3 months
Phase II: Increase in fetal hemoglobin (HbF) as measured by hemoglobin electrophoresis | Baseline, 6 months, 1 year

SECONDARY OUTCOMES:
Phase II: Measures of adherence to HU | Baseline, 6 months, 1 year
  For patients prescribed HU, clinical research coordinators will assess HU prescription refills from pill counts, pharmacy records, and self-report at baseline, 6 months, and 1 year. Patient navigators will regularly assess their patients' HU adherence by conducting pill counts at home visits.
Phase II: Percent of patients achieving either maximum tolerated dose (MTD) or maximum dose | Baseline, 6 months, 1 year
  Maximum tolerated dose (MTD) is the daily single oral dose that can be maintained for at least 16 weeks without toxicity (< 3 x l09 neutrophils/L, <100 x l09 platelets/L, < 125 x l09 reticulocytes/L, 20% drop in [Hb] or an absolute value of <4.5 g/dL, 50% rise in creatinine or absolute increase of >0.4 mg/dL, 100% rise in ALT,GI disturbance, or rash or hair loss not attributable to other causes). Maximum dose is 35 mg/kg.
Phase II: Number of emergency department and hospital visits | Baseline, 6 months, 1 year
Phase II: Mean corpuscular volume | Baseline, 6 months, 1 year
Phase II: Total hemoglobin | Baseline, 6 months, 1 year
Phase II: White blood cell count | Baseline, 6 months, 1 year
Phase II: Reticulocyte count | Baseline, 6 months, 1 year
Phase II: Quality of life measures | Baseline, 6 months, 1 year
  Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me), Patient Reported Outcomes Measurement Information System (PROMIS)
Phase II: Patient activation measures | Baseline, 6 months, 1 year
  Patient Activation Measure
Phase II: Patient knowledge measures | 1 year
  Assessment of Sickle Cell Knowledge - University of Florida (UF-ASCK) (unpublished)
Phase II: Health care knowledge and skills, self-efficacy, sickle cell stress measures | Baseline, 6 months, 1 year
  Sickle Cell Transition intervention Program (TIP) Survey (non-validated)
Phase II: Social support measures | Baseline, 6 months, 1 year
  Sickle Cell Transition intervention Program (TIP) Survey (non-validated) and Multidimensional Scale of Perceived Social Support
Phase II: Coping strategies | Baseline, 6 months, 1 year
  Coping Strategies Questionnaire for SCD
Phase II: Associated pain conditions and comorbidities | Baseline, 6 months, 1 year
  Chart Review, Self Report and Surveys: Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me), Patient Reported Outcomes Measurement Information System (PROMIS)
Phase II: Blood transfusion measures (if applicable) | 6 months, 1 year
  Chart review
Phase II: Patient Navigator Satisfaction (if applicable) | 1 year
  Patient Navigator Satisfaction Surveys, 12 month follow up, Patient Study Experience Review for Patient Navigators

CONTACTS AND LOCATIONS:
Overall Officials: Wally R Smith, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClish D, Okhomina V, Pascale A, Valrie C, Sisler I, Villella A, Smith W. Vaso-occlusive crisis pain intensity, frequency, and duration: which best correlates with health-related quality of life in adolescents and adults with sickle cell disease? Pain. 2024 Jan 1;165(1):135-143. doi: 10.1097/j.pain.0000000000003011. Epub 2023 Aug 11. PMID 37578485
- [Derived] Smith WR, Valrie C, Sisler I. Structural Racism and Impact on Sickle Cell Disease: Sickle Cell Lives Matter. Hematol Oncol Clin North Am. 2022 Dec;36(6):1063-1076. doi: 10.1016/j.hoc.2022.08.008. PMID 36400531
- [Derived] Sisler I, McClish DK, Valrie C, Villella A, Smith WR. Satisfaction and access to care for adults and adolescents with sickle cell disease: ASCQ-Me quality of care and the SHIP-HU study. Pediatr Blood Cancer. 2022 Dec;69(12):e29948. doi: 10.1002/pbc.29948. Epub 2022 Sep 24. PMID 36151945

DOCUMENTS (1):
  • Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT02197845/ICF_000.pdf